CLINICAL TRIAL: NCT00315146
Title: Optimizing Body Composition for Function in Older Adults (OPTIMA) - A Pepper Pilot Study
Brief Title: Optimizing Body Composition for Function in Older Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Takeda Pharmaceuticals North America, Inc. (Industry); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: BG06-051; P30AG021332 (NIH)
Record Dates: First submitted 2006-04-13; First posted 2006-04-17 (Estimated); Results first posted 2014-12-19 (Estimated); Last update posted 2018-08-28 (Actual); Status verified 2018-07

CONDITIONS: Obesity; Overweight With Indications for Weight Loss
Keywords: Body Composition; Sarcopenia; Weight loss trials; Intervention studies; Elderly
MeSH Terms: conditions — Obesity; Sarcopenia | interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Hypocaloric diet (and placebo) (Placebo Comparator)
  Interventions: Behavioral: Hypocaloric diet; Drug: Placebo
- Hypocaloric diet, resist. training to maximize power, placebo (Active Comparator)
  Interventions: Behavioral: Resistance exercise training to maximize muscle power; Behavioral: Hypocaloric diet; Drug: Placebo
- Hypocaloric diet and a PPAR- γ agonist (pioglitazone/Actos™) (Active Comparator)
  Interventions: Drug: Pioglitazone; Behavioral: Hypocaloric diet
- Hypocaloric diet,resistance training, pioglitazone/Actos™ (Active Comparator)
  Interventions: Drug: Pioglitazone; Behavioral: Resistance exercise training to maximize muscle power; Behavioral: Hypocaloric diet

INTERVENTIONS:
Drug: Pioglitazone
  Arms: Hypocaloric diet and a PPAR- γ agonist (pioglitazone/Actos™); Hypocaloric diet,resistance training, pioglitazone/Actos™
Behavioral: Resistance exercise training to maximize muscle power
  Arms: Hypocaloric diet, resist. training to maximize power, placebo; Hypocaloric diet,resistance training, pioglitazone/Actos™
Behavioral: Hypocaloric diet
Drug: Placebo
  Arms: Hypocaloric diet (and placebo); Hypocaloric diet, resist. training to maximize power, placebo

SUMMARY:
The purpose of this pilot study is to compare two strategies intended to improve the health of overweight older adults by improving body composition. One strategy, resistance training, is designed to preserve skeletal muscle mass. The other strategy, the use of a PPAR-γ agonist, is designed to enhance the loss of fat from visceral and skeletal depots. These strategies will be used in conjunction with a hypocaloric diet and will be compared to a hypocaloric diet alone to determine if either of these strategies are superior in reducing visceral fat and preserving muscle mass.

DETAILED DESCRIPTION:
In this pilot we propose to recruit 88 older (65 - 79 yrs) men (n=48) and women (n=40) at risk for disability and with indications for weight loss according to NIH guidelines. All will be enrolled in a dietary intervention designed to generate a caloric deficit of 500 kcal/day for a 4 month period. All will receive supplemental vitamin D and calcium. These participants will be randomized into one of 4 groups:

Group 1 - Hypocaloric diet (and placebo) Group 2 - Hypocaloric diet and resistance training designed to maximize muscular power (and placebo) Group 3 - Hypocaloric diet and a PPAR- γ agonist (pioglitazone/Actos™) Group 4 - Hypocaloric diet and resistance training and pioglitazone/Actos™

The specific aims of the pilot are:

1. In both men and women, to determine whether randomization to resistance exercise is associated with an increased retention of appendicular non-bone lean mass compared to those not undergoing power training.
2. In both men and women, to determine whether randomization to the pioglitazone group is associated with an increased loss of visceral adiposity relative to randomization to the non-pioglitazone group.
3. Assess the feasibility of the recruitment, assessment and intervention strategies
4. To estimate adherence to the weight loss, exercise training, and drug interventions;
5. In this population, to determine measurement characteristics of the functional outcomes that will be considered as primary end-points of the larger study.
6. To obtain pilot data on a subset of participants to determine the feasibility, acceptability and measurement characteristics of muscle samples (biopsies) to quantify intramyocellular lipid in this study population.

ELIGIBILITY:
Inclusion Criteria:

* Weight Stable, Indication for weight loss per NIH guidelines, Performance on the short physical performance battery score 3-10

Exclusion Criteria:

* Diabetes, weight > 136 kg, Medical condition that limits exercise participation, Congestive heart failure, abnormal kidney function, higher ALT than normal, currently involved in a weight loss or exercise program, current smoking, alcohol or drug abuse, taking anti-inflammatory steroids, taking protein supplements, taking PPAR-gamma agonist, edema, anemia

Ages: 65 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 88 (Actual)
Dates: Start 2006-04; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen B Kritchevsky, PhD, Principal Investigator — Sticht Center on Aging, Wake Forest University School of Medicine
Locations (1):
- Sticht Center on Aging, Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Starting in April 2006,144 participants underwent a medical screening. After further exclusion (n = 47) and declining to participate (n = 9), 88 participants (48 men, 40 women) were randomized to one of the four treatment groups.
Groups:
- Hypocaloric Weight Loss Only: Two meal replacements per day (bars and shakes) were provided to all participants (containing ~220 kcal with 7-10 g protein, 33-46 g carbohydrates, and 1.5-5 g fat with 2-5 g of fiber). For the third meal, a weekly menu plan with recipes was given to the participants. This meal was composed of traditional foods, was low in fat, high in vegetables but allowed for individual preferences, and provided 500-750 kcal. In addition, up to three snacks (~100 kcal each) were allowed each day. The macronutrient goal for each individual was ~55-60% carbohydrates, ~15% protein, and ~25% fat.
- Hypocaloric Weight Loss + Pioglitazone: Two meal replacements per day (bars and shakes) were provided to all participants (containing ~220 kcal with 7-10 g protein, 33-46 g carbohydrates, and 1.5-5 g fat with 2-5 g of fiber). For the third meal, a weekly menu plan with recipes was given to the participants. This meal was composed of traditional foods, was low in fat, high in vegetables but allowed for individual preferences, and provided 500-750 kcal. In addition, up to three snacks (~100 kcal each) were allowed each day.
  Pioglitazone was given an initial 15 mg/day dose. Participants were assessed for side effects after 3 weeks, but none were reported. Therefore, after 3 weeks, the dose was increased to 30 mg/day for the remainder of the study for all participants randomized to receive pioglitazone. In order to understand the potential effects of changes in body composition independent of drug effects, a 1-week wash-out period preceded the follow-up outcome assessment.
- Hypocaloric Weight-loss +Resistance Training: Two meal replacements per day (bars and shakes) were provided to all participants (containing ~220 kcal with 7-10 g protein, 33-46 g carbohydrates, and 1.5-5 g fat with 2-5 g of fiber). For the third meal, a weekly menu plan with recipes was given to the participants. This meal was composed of traditional foods, was low in fat, high in vegetables but allowed for individual preferences, and provided 500-750 kcal. In addition, up to three snacks (~100 kcal each) were allowed each day.
  The goal of the resistance training program was to increase strength and muscle mass in the major muscle groups of the body, while also improving muscle power in the lower extremity. Participants randomized to the resistance training exercised 3 days/week. Participants warmed-up by walking or cycling for 3-5 min at a slow pace followed by 5 min of large muscle flexibility exercises targeting the major muscle groups of the body. Training sessions ended with a cool-down session of light stretching.
- Hypocaloric Weight Loss + Resistance Training + Pioglitazone: Two meal replacements per day (bars and shakes) were provided to all participants (containing ~220 kcal with 7-10 g protein, 33-46 g carbohydrates, and 1.5-5 g fat with 2-5 g of fiber). For the third meal, a weekly menu plan with recipes was given to the participants.
  The goal of the resistance training program was to increase strength and muscle mass in the major muscle groups of the body, while also improving muscle power in the lower extremity. Participants randomized to the resistance training exercised 3 days/week. Participants warmed-up by walking or cycling for 3-5 min at a slow pace followed by 5 min of large muscle flexibility exercises targeting the major muscle groups of the body.
  Pioglitazone was given an initial 15 mg/day dose. Participants were assessed for side effects after 3 weeks. Therefore, after 3 weeks, the dose was increased to 30 mg/day for the remainder of the study for all participants randomized to receive pioglitazone.
Period: Overall Study
Arm/Group | Hypocaloric Weight Loss Only | Hypocaloric Weight Loss + Pioglitazone | Hypocaloric Weight-loss +Resistance Training | Hypocaloric Weight Loss + Resistance Training + Pioglitazone
Started | 22 | 22 | 22 | 22
Completed | 20 | 19 | 20 | 22
Not Completed | 2 | 3 | 2 | 0

BASELINE CHARACTERISTICS:
Population: These numbers match the number of people who STARTED in each group in the flow module.
Groups:
- Total: Total of all reporting groups
Arm/Group | Hypocaloric Weight Loss Only | Hypocaloric Weight Loss + Pioglitazone | Hypocaloric Weight-loss +Resistance Training | Hypocaloric Weight Loss + Resistance Training + Pioglitazone | Total
Number analyzed (Participants) | 22 | 22 | 22 | 22 | 88
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 22 | 22 | 22 | 22 | 88
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.0 (3.9) | 70.4 (3.5) | 71.0 (4.3) | 69.9 (2.7) | 70.6 (3.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 10 | 10 | 40
  Male | 12 | 12 | 12 | 12 | 48
Region of Enrollment [Number; unit: participants]
  United States | 22 | 22 | 22 | 22 | 88

OUTCOME MEASURES:

1. Primary Outcome: Appendicular Non-bone Lean Mass
Description: Change in Appendicular Non-bone Lean Mass
Time Frame: Baseline visit (pre intervention) and 4month follow up (post intervention)
Measure: Least Squares Mean (95% Confidence Interval); unit: kg
Arm/Group | Hypocaloric Weight Loss Only | Hypocaloric Weight Loss + Pioglitazone | Hypocaloric Weight-loss +Resistance Training | Hypocaloric Weight Loss + Resistance Training + Pioglitazone
Number analyzed (Participants) | 20 | 19 | 20 | 22
kg | -2.53 [-3.34 to -1.72] | -2.49 [-3.32 to -1.66] | -2.04 [-2.86 to -1.23] | -1.45 [-2.22 to -0.67]

2. Secondary Outcome: Lean Body Mass
Time Frame: Baseline visit (pre intervention) and 4month follow up (post intervention)
Measure: Least Squares Mean (95% Confidence Interval); unit: kg
Groups:
- Hypocaloric Diet (and Placebo): Hypocaloric diet
  Placebo
- Hypocaloric Diet, Resist. Training to Maximize Power, Placebo: Resistance exercise training to maximize muscle power
  Hypocaloric diet
  Placebo
- Hypocaloric Diet and a PPAR- γ Agonist (Pioglitazone/Actos™): Pioglitazone
  Hypocaloric diet
- Hypocaloric Diet,Resistance Training, Pioglitazone/Actos™: Pioglitazone
  Resistance exercise training to maximize muscle power
  Hypocaloric diet
Arm/Group | Hypocaloric Diet (and Placebo) | Hypocaloric Diet, Resist. Training to Maximize Power, Placebo | Hypocaloric Diet and a PPAR- γ Agonist (Pioglitazone/Actos™) | Hypocaloric Diet,Resistance Training, Pioglitazone/Actos™
Number analyzed (Participants) | 20 | 20 | 19 | 22
kg | -2.55 [-4.31 to -0.79] | -1.89 [-3.99 to -.021] | -2.38 [-4.48 to -0.28] | -1.65 [-3.67 to 0.37]

ADVERSE EVENTS:
Arm/Group | Hypocaloric Weight Loss Only | Hypocaloric Weight Loss + Pioglitazone | Hypocaloric Weight-loss +Resistance Training | Hypocaloric Weight Loss + Resistance Training + Pioglitazone
Serious Adverse Events (participants affected / at risk) | 3/22 | 0/22 | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 0/22 | 0/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hypocaloric Weight Loss Only (N=22) | Hypocaloric Weight Loss + Pioglitazone (N=22) | Hypocaloric Weight-loss +Resistance Training (N=22) | Hypocaloric Weight Loss + Resistance Training + Pioglitazone (N=22)
Hospitalization for DVT (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hospitalization for brain tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fainted during muscle biopsy procedure (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes